CLINICAL TRIAL: NCT06209333
Title: Effect of Bladder Training and Pelvic Floor Exercise Training on Urinary Symptoms and Quality of Life in Patients With Overactive Bladder Syndrome
Brief Title: Effect of BT and PFET on Urinary Symptoms and Quality of Life in Patients With OABS
Acronym: OABS/BT/PFET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceren Gursen, Associate professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-23003
Record Dates: First submitted 2023-09-18; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Overactive Bladder Syndrome (OABS)
Keywords: pelvic floor exercise; bladder training; standard patient education; botulinum toxin-A; BTx-A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pelvic physiotherapy (Experimental)
  Interventions: Other: bladder training; Other: pelvic floor exercise
- standard patient education (Active Comparator)
  Interventions: Other: Standard Patient Education

INTERVENTIONS:
Other: Standard Patient Education — Standard Patient Education will take approximately 20 minutes. Within the scope of standard patient education, some recommendations will be made to the patient to lose weight, drink sufficient water, avoid consuming caffeinated foods and beverages, acidic/carbonated or alcoholic beverages, spicy/acidic foods, and quit smoking. Patients will be evaluated on the day they receive standard patient training (before receiving this training) and 10 weeks after the training.
  Arms: standard patient education
Other: bladder training — Interval urination in bladder training in bladder training will be determined according to the bladder diaries filled in by the patients. If the patient is able to do it, bladder education will be improved by increasing the interval urination in bladder training. A total of 5 sessions of bladder training will be applied to patients, the first session of which will be face-to-face. Within the scope of Bladder Training, the patient will be given information about bladder, pelvic floor, incontinence and relaxation techniques. The patient will be asked to fill out a 3-day bladder diary before starting bladder training, and an appropriate progressive timed voiding program will be drawn according to the bladder diaries, and the patient will be given a training brochure to implement this program.
  Arms: pelvic physiotherapy
Other: pelvic floor exercise — This training will take between 45 and 60 minutes.Within the scope of exercise training, patients will be taught 3 types of contractions: maximal (fast), slow and submaximal contractions. The patient will be asked to continue the maximum and submaximal contraction for 1-2 seconds, and to continue the Deceleration contraction for 3-10 seconds. These contractions will be performed in different positions such as supine, lying on the side, sitting, crawling, squatting and standing, specifically for the pelvic floor November muscle strength of the patient. These exercises will be performed every day and each type of contraction (maximal, slow and submaximal contraction) will be performed 8-12 repetitions, 3 sets per day. Progress will be achieved with follow-ups.
  Arms: pelvic physiotherapy

SUMMARY:
The aim of this study was to examine the effects of bladder training and pelvic floor exercise training programs given in addition to Botulinum Toxin-A (BTx-A) application on urinary symptoms and quality of life in patients with Overactive Bladder Syndrome (AAMS) who do not respond to conservative treatments.

Individuals who meet the criteria for inclusion in the study and agree to participate in the study will be divided into 2 separate research branches.The patients to be included in the study will be divided into two groups as "Group 1=Botox + physiotherapy " or "Group 2=Botox group ". In addition to the BTx-A application, bladder training and pelvic floor exercise training will be applied to patients in the first group, while standard patient training will be provided to patients in the second group.

Severity of urinary symptoms, quality of life and subjective perception of improvement Before BTx-A application, 2 weeks and 12 weeks after BTX-A application, International Incontinence Consultation Questionnaire - Women's Lower Urinary Tract Symptoms (ICIQ-FLUTS), 1-hour ped test, International Incontinence Consultation- Lower Urinary Tract Symptoms Quality of Life Scale (ICIQ-LUTS) and Global Perception of Improvement will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 (those with a Mini Mental Test score of 24 and above for individuals over the age of 65),
* Who has Non-Neurogenic Overactive Bladder Syndrome,
* Patients who received Routine Botulinum Toxin-A administration because they did not respond to conservative treatment,
* Patients who volunteer to participate in the study will be included.

Exclusion Criteria:

* Patients with Neurogenic Overactive Bladder Syndrome,
* Pregnant Women,
* Lack of cooperation in evaluation and/or treatment and lack of literacy status,
* Patients with urogynocological/anatomical abnormalities,
* Patients receiving pelvic radiation therapy,
* Patients with psychiatric or neurogenic disorders and
* Patients who have not given consent to the study and do not have an informed consent form (BGOF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
International Incontinence Consultation Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) | the change in the symptoms of the lower urinary tract from the beginning to the end of 12 weeks and the effects of symptoms on quality of life
  Storage symptoms are scored as 0-16 points, urination symptoms are scored as 0-12, incontinence symptoms are scored as 0-20 points.
  The effect of the patient's symptoms on their daily activities has 5 options, including "0-Never", "4-Always".The highest possible score is 48. A higher score means a worse outcome.
International Incontinence Consultation Questionnaire - Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) | the change in the symptoms of the lower urinary tract from the beginning to the end of 12 weeks and the effects of symptoms on quality of life
  This scale aims to evaluate male lower urinary tract symptoms in the last 4 weeks and the effects of symptoms on quality of life with 13 questions.
  The effect of the patient's symptoms on their daily activities has 5 options, including "0-Never", "4-Always".The highest possible score is 52. A higher score means a worse outcome.

SECONDARY OUTCOMES:
International Incontinence Consultation Bladder Diary (ICIQ-Bladder Diary): | change in the severity of urinary incontinence from the beginning to the end of 12 weeks
  ICIQ-Bladder Diary is a volume-frequency chart that allows patients to record the frequency of urination, the volume of mixing and fluid intake (quantity, duration and type), bladder sensation and pad use at each time.
1-Hour Ped Test | change in the severity of urinary incontinence from the beginning to the end of 12 weeks
  Just before this test, the patient is asked to empty his bladder and put the pad, the weight of which is known in advance, in his clothes.
  Then, the patient is asked to do 500 mL of oral hydration while sitting for 15 minutes. the time is completed with other activities.
  60. the pad is taken from the patient per minute. During this time, the weight difference on the pad is measured and the test is interpreted according to the difference.
International Incontinence Consultation- Lower Urinary Tract Symptoms Quality of Life Scale (ICIQ-LUTS): | Change in quality of life from baseline at 12 weeks
  Quality of life will be evaluated by the International Incontinence Consultation- Lower Urinary Tract Symptoms Quality of Life Scale (ICIQ-LUTS). This scale consists of 20 questions that evaluate different sub-areas of quality of life (work life, daily life, travel and sexuality).The highest possible score is 76. A higher score means a worse outcome.
Global Perception of Improvement Scale | Change from baseline patient global change at 12 weeks
  The Global Perception of Improvement Scale, the perception of changes in patients' complaints related to overactive bladder symptoms after the study compared to the beginning of the study, will be evaluated by the Global Perception of Improvement Scale, which is a 7-item scale (1-I am much better, 7-much worse). A higher score means a worse outcome.
Compliance with Standard Patient Education | compliance with Standard Patient Education at the end of 12 weeks
  It will be evaluated with a Visual Analog Scale. The Visual Analog Scale (VAS) is a horizontal line of 0-10 cm that expresses that it does not fit education at all at one end and that it adapts to patient education to the maximum extent at the other end. A higher score means better fit.
Compliance with Bladder Training | Compliance with Bladder Training at the end of 12 weeks
  It will be evaluated with a Visual Analog Scale. 12. at the end of the week, they will be asked to mark on the VAS how much they have implemented this training throughout the study.
Compliance with Pelvic Floor Exercise Training | Compliance with Pelvic Floor Exercise Training at the end of 12 weeks
  It will be evaluated with exercise diaries.

CONTACTS AND LOCATIONS:
Locations (1):
- Aslı Aslan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The Overactive Bladder: From Basic Science to Clinical Management Consensus Conference. Proceedings. London, England, June 29, 1997. Urology. 1997 Dec;50(6A Suppl):1-114. No abstract available. PMID 9446279
- [Background] Orasanu B, Mahajan ST. The use of botulinum toxin for the treatment of overactive bladder syndrome. Indian J Urol. 2013 Jan;29(1):2-11. doi: 10.4103/0970-1591.109975. PMID 23671356
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Mertoglu O, Ucer O, Ceylan Y, Bozkurt O, Gunlusoy B, Albaz AC, Demir O; Aegean Study Group of Society of Urological Surgery. Reliability and Validity of the Turkish Language Version of the International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms. Int Neurourol J. 2016 Jun;20(2):159-63. doi: 10.5213/inj.1630460.230. Epub 2016 Jun 24. PMID 27377949
- [Background] Shen L, Hou L, Li B, Jin X, Han F, Wang Y. Translation of the ICIQ-bladder diary and its validation among Chinese females with lower urinary tract symptoms. Int Urogynecol J. 2020 Dec;31(12):2535-2542. doi: 10.1007/s00192-020-04339-9. Epub 2020 May 28. PMID 32468173
- [Background] Castellani D, Saldutto P, Galica V, Pace G, Biferi D, Paradiso Galatioto G, Vicentini C. Low-Dose Intravaginal Estriol and Pelvic Floor Rehabilitation in Post-Menopausal Stress Urinary Incontinence. Urol Int. 2015;95(4):417-21. doi: 10.1159/000381989. Epub 2015 May 30. PMID 26043913
- [Background] Ptak M, Ciecwiez S, Brodowska A, Starczewski A, Nawrocka-Rutkowska J, Diaz-Mohedo E, Rotter I. The Effect of Pelvic Floor Muscles Exercise on Quality of Life in Women with Stress Urinary Incontinence and Its Relationship with Vaginal Deliveries: A Randomized Trial. Biomed Res Int. 2019 Jan 6;2019:5321864. doi: 10.1155/2019/5321864. eCollection 2019. PMID 30723739